CLINICAL TRIAL: NCT03823989
Title: An Open-label, Phase 1b Study of Intravenously Administered Pegylated Liposomal Mitomycin C Lipid-based Prodrug (PROMITIL) in Combination With External Beam Radiotherapy in Patients With Advanced Cancer Requiring Palliative Radiotherapy
Brief Title: Intravenously Administered Liposomal PROMITIL in Combination With External Beam Radiotherapy in Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lipomedix Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LIPORAD-2018
Record Dates: First submitted 2019-01-22; First posted 2019-01-31 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Cancer; Solid Tumor; Metastatic Disease
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: dose-escalation study will begin with a dose of 1.25 mg/kg, to be followed by an increase to 1.5 mg/kg PROMITIL and a further increase 1.8 mg/kg in the absence of DLTs after two treatment cycles, with an interluding 10-fraction course of radiotherapy. Upon completion of two treatment cycles, with ≤1 incident of DLTs in Cohort 2, a third confirmatory cohort (n=6) will be recruited and will be treated with the same dose as that administered to Cohort 2
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Promitil 1.25 mg/kg (Experimental): Two treatment cycles, intravenous infusion of Promitil at a dosage of 1.25 mg/kg delivered at 21 days interval and a 10-fraction course of EBR (3 Gy/fraction), initiated 1-3 days after the first PROMITIL dose and completed within a 2-week period.
  Interventions: Drug: Promitil; Radiation: EBR
- Promitil 1.5 mg/kg (Experimental): Two treatment cycles, intravenous infusion of Promitil at a dosage of 1.5 mg/kg delivered at 21 days interval and a 10-fraction course of EBR (3 Gy/fraction), initiated 1-3 days after the first PROMITIL dose and completed within a 2-week period.
  Interventions: Drug: Promitil; Radiation: EBR
- Promitil 1.8 mg/kg (Experimental): two treatment cycles, intravenous infusion of Promitil at a dosage of 1.8 mg/kg delivered at 21 days interval (confirmatory cohort) and a 10-fraction course of EBR (3 Gy/fraction), initiated 1-3 days after the first PROMITIL dose and completed within a 2-week period.
  Interventions: Drug: Promitil; Radiation: EBR

INTERVENTIONS:
Drug: Promitil — The first 6 patients recruited to the study will receive 1.25 mg/kg PROMITIL. If no dose-limiting toxicities (DLTs) are recorded by day 43 of the study, the second cohort of 6 patients will begin treatment at a dose level of 1.5 mg/kg PROMITIL. Upon completion of two treatment cycles, with ≤1 incident of DLTs in Cohort 2, a third cohort (n=6) will be recruited and will be treated with a dose level of 1.8 mg/kg.
  Other Names: Pegylated Liposomal Mitomycin-C Lipid-based Prodrug
Radiation: EBR — A 10-fraction course of EBR (3 Gy/fraction), initiated 1-3 days after the first PROMITIL dose and completed within a 2-week period.
  Other Names: external beam radiotherapy

SUMMARY:
This will be a multi-center, open-label, single-arm, prospective study, in which up to 18 adult patients requiring radiotherapy for metastatic disease or for an inoperable primary tumor with no definitive curative treatment option, will undergo a combination treatment of intravenously (IV) delivered PROMITIL and standard of care radiotherapy. The treatment regimen will involve administration of two PROMITIL doses, delivered at a 21-day interval, and a course of EBR (type of RT according to investigator's preference), initiated 1-3 days after the first PROMITIL dose and completed within a 2-week period. EBR will consist of no more than 10 fractions delivered within 2 weeks as conventionally fractionated RT, or SBRT. Treatment safety will be assessed on a weekly basis throughout the two 21-day treatment courses (42 days) and throughout the follow-up period (up to Day 127). AEs will only be logged until 6 weeks after the last PROMITIL dose (up until Day 64). Disease status will be reevaluated between days 43-50 of the study, and every 6 weeks thereafter (Days 85 and 127±7 days). In addition, following completion of the treatment schedule, all patients will be followed up by phone every 12 weeks, until either death, disease progression (PD), withdrawn consent or trial cut-off date, i.e., for up to 2 years after patient accrual to study, (whichever occurs first). The following anticancer agents will NOT be allowed during the screening period, 6-week treatment period and until first disease reevaluation: cytotoxic agents, non-cytotoxic myelosuppressive agents (CDK 4/6 inibitiors, PARP inhibitors, m-TORS inhibitors and tyrosine kinase-inhibitors). Treatment with hormonal agents, monoclonal antibodies (anti-EGFr, anti-Her2, anti-VEGF and VEGFr, anti-PD1, anti-PDL1) and bisphosphonates can be continued during the study.

DETAILED DESCRIPTION:
As combination with radiotherapy is expected to provide an additive or synergistic effect, the current dose-escalation study will begin with a dose of 1.25 mg/kg, to be followed by an increase (1.5 mg/kg) in Cohort 2 and a further increase 1.8 mg/kg in Cohort 3 in the absence of DLTs after two treatment cycles, with an interluding 10-fraction course of radiotherapy.

PROMITIL will be intravenously delivered on Day 1 of each of the two 21-day cycles.

Cohort 1: The first 6 patients recruited to the study will receive 1.25 mg/kg PROMITIL.

Cohort 2: If no dose-limiting toxicities (DLTs) are recorded by day 43 of the study, the second cohort of 6 patients will begin treatment at a dose level of 1.5 mg/kg PROMITIL. However, if 1 DLT is recorded, the second cohort of 6 patients will receive the same dose of 1.25 mg/kg PROMITIL. If 2 DLTs are recorded in Cohort 1, the second cohort of 6 patients will receive 1.0 mg/kg PROMITIL.

Cohort 3: If no dose-limiting toxicities (DLTs) are recorded by day 43 of the study of the first 3 patients of Cohort 2, a third cohort will enroll 6 patients to receive treatment at a dose level of 1.8 mg/kg PROMITIL. If none or 1 DLT is recorded, the dose of 1.8 mg/kg will be cleared as recommended dose for phase 2. If 2 DLT are recorded, the study will be terminated as soon as the 2nd DLT is recorded, and the prior dose level of 1.5 mg/kg will be cleared as recommended dose for phase 2

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed recurrent and/or metastatic, cancer, with at least one measurable lesion (≤10 cm diameter) on file, and with no definitive curative treatment option.
2. A ≥21-day treatment-free interval from last chemotherapeutic treatment (including cytotoxic or non-cytotoxic myelosuppressive agents), and ≥14-day treatment-free interval from biological therapies consisting of CDK 4/6 inibitiors, PARP inhibitors, m-TOR inhibitors Hormonal therapies including LH-RH analogs or anagonists, tamoxifen, aromatase inhibitors, bicalutamide, aboraterone, corticosteroids, or enzalutamide may be continued uninterruptedly.
3. No prior intravenous treatment with mitomycin-C either alone or in combination
4. No prior extensive radiotherapy (e.g., whole pelvis, or greater than 50% of neuroaxis, whole abdomen, whole body or half-body) or bone marrow transplantation with high dose chemotherapy.
5. No prior radiotherapy to the same anatomic site aimed for radiotherapy.
6. Age ≥18years
7. BMI: 18-36
8. ECOG Performance Status ≤ 2
9. Estimated life expectancy of at least 3 months
10. Adequate bone marrow function (an absolute neutrophil count ≥1500/mm3, hemoglobin ≥9.5 g/dl, and a platelet count ≥100,000/mm3);
11. Adequate liver function (serum bilirubin ≤2.0 mg/100 ml; alanine aminotransferase ≤3× ULN, albumin ≥34g/L)
12. Adequate renal function (serum creatinine ≤1.5 mg/100 ml or creatinine clearance ≥40 ml/min/1.73m2)
13. Women of child-bearing potential practicing an acceptable method of birth control.
14. Understanding of study procedures and willingness to comply for the entire length of the study and to provide written informed consent

Exclusion Criteria:

1. Known hypersensitivity to the study drug or to any of its components
2. Prior intravenous treatment with mitomycin C
3. Patients requiring whole-brain irradiation
4. Patients requiring re-irradiation of the same tumor/anatomical site.
5. CHF (NYHA = Class IV)
6. Severe COPD or Stage ≥3 severe emphysema with FEV1 between 30 and 50 percent of normal
7. Chronic liver disease or cirrhosis with Child-Pugh Class C score
8. Any other severe concurrent disease which in the judgment of the investigator would make the subject unsuitable for entry into this study
9. History of human immunodeficiency virus (HIV) infection
10. History of chronic active hepatitis including subjects who are carriers of hepatitis B virus (HBV) or hepatitis C virus (HCV), unless adequately treated and shown to be serum virus-free.
11. Presence of uncontrolled infection.
12. Evidence of active bleeding or bleeding diathesis
13. Pregnant or lactating
14. Treatment with other investigational drugs within <21 days of start of day 1 of study drug.
15. Uncontrolled ascites (defined as 2 or more palliative taps in the last 21 days before screening).

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) of Promitil in combination with external beam radiotherapy (EBR) | 6 weeks
  Report of Dose limiting toxicity
Incidence of Treatment-Emergent Adverse Events | 6 weeks
  Incidence all Adverse events of Promitil in combination with external beam radiotherapy (EBR)
To evaluate the response rate to PROMITIL in combination with external beam radiotherapy (EBR) | 7 weeks
  Local disease control in irradiated tumor areas at first reevaluation (Day 43-50), defined as rate of complete response [CR], partial response [PR] and stable disease [SD], as per RECIST 1.1 criteria

SECONDARY OUTCOMES:
Duration of response of the irradiated tumor site | 18 weeks
  Duration of response (in weeks) of the irradiated tumor site, from first evidence of response (Stable disease or better) to confirmed Progression disease (as per RECIST 1.1 criteria)
Progression-free survival (PFS) | 18 weeks
  Progression-free survival (PFS) (in weeks), from day of first dose of PROMITIL until confirmed Progression disease (as per RECIST 1.1 criteria)
Overall survival | 34 weeks
  Overall survival (in weeks), from day of first dose of PROMITIL to death of any cause
Plasma MLP level after Promitil infusion | 6 weeks (2 cycles of treatment)
  Plasma MLP levels before and after (1 h and 24 h) each PROMITIL dose

CONTACTS AND LOCATIONS:
Overall Officials: Adi Levy, MD, Principal Investigator — Hadassah Medical Organization; Eli Sapir, MD, Study Director — Assuta Medical Center
Locations (3):
- Israel (3):
  - Assuta Ashdod, Ashdod
  - Hadassah Medical Center, Jerusalem
  - Assuta Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No
The PI and the sponsor have still to discuss what will be the plan to share IPD

REFERENCES:
- [Background] Tian X, Warner SB, Wagner KT, Caster JM, Zhang T, Ohana P, Gabizon AA, Wang AZ. Preclinical Evaluation of Promitil, a Radiation-Responsive Liposomal Formulation of Mitomycin C Prodrug, in Chemoradiotherapy. Int J Radiat Oncol Biol Phys. 2016 Nov 1;96(3):547-55. doi: 10.1016/j.ijrobp.2016.06.2457. Epub 2016 Jul 1. PMID 27681751
- [Background] Tahover E, Bar-Shalom R, Sapir E, Pfeffer R, Nemirovsky I, Turner Y, Gips M, Ohana P, Corn BW, Wang AZ, Gabizon AA. Chemo-Radiotherapy of Oligometastases of Colorectal Cancer With Pegylated Liposomal Mitomycin-C Prodrug (Promitil): Mechanistic Basis and Preliminary Clinical Experience. Front Oncol. 2018 Nov 26;8:544. doi: 10.3389/fonc.2018.00544. eCollection 2018. PMID 30534533